CLINICAL TRIAL: NCT03896607
Title: Prospective Study: Shear-Wave Elastography of the Liver and the Spleen in Adult Patients With Gaucher's Disease
Brief Title: Liver and the Spleen Stifness in Adult Patients With Gaucher's Disease Using Ultrasound Shear Wave Elastography
Status: Terminated | Type: Observational
Why Stopped: study has ended due to internal changes
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Ziv Neeman, Head of Radiology department, HaEmek Medical Center, Israel
Other Study IDs: 0135-18-EMC
Record Dates: First submitted 2019-03-17; First posted 2019-04-01 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Gaucher Disease; Liver Fibrosis; Spleen; Fibrosis
Keywords: shear wave elastography
MeSH Terms: conditions — Gaucher Disease; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigated cohort will examine liver and spleen fibrosis in patients with Gaucher Disease(GD) by using Shear Wave Elastography- SWE to evaluation fibrosis of the tissue and to check the correlation of fibrosis with the biomarkers of disease severity.

DETAILED DESCRIPTION:
To assess liver and spleen stiffness measurement using Shear Wave Elastography-SWE and evaluate liver and spleen fibrosis in patients with Gaucher Disease. To compare the elastography with the biomarkers that taken at the GD haematology clinic and to check the correlation with severity of liver and spleen fibrosis.

SWE is a safe with diagnostic accuracy regarding the liver (& Spleen) fibrosis. Estimating spleen fibrosis is an innovative approach in liver disease and Gaucher.

The evaluation of fibrosis with this relatively new and safe method could avoid complications and invasive procedure in GD patients .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Gaucher disease over the age of 18 years.
2. Patients able to sign informed consent form.
3. Women are not pregnant.
4. Patients who read and understood the contents of the consent form and gave their written consent to participate in the study.

Exclusion Criteria:

1. Participants under the age of 18.
2. Pregnant women.
3. Participants are unable to sign an informed consent form.
4. Participants with known liver disease not associated with Gaucher disease such as liver cirrhosis, patients with HBV, HBC or liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient with Gaucher disease.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Shear Wave Elastography of liver to asses liver fibrosis in Gaucher disease patients. | 0-2 hours
  Shear wave elastography(SWE),an ultrasound imaging technique that can produce 2D and 3D images and quantified measurements of tissue stiffness noninvasively. SWE obtained from the right liver lobe for staging liver fibrosis according to Metavir Fibrosis Score with sensitivity86%-98% and specificity 90%-93%. SWE well corelated with Metavir Fibrosis Score which is system used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy. The biomarkers of disease severity will be correlated to METAVIR score. METAVIR score(F0-F4) ,Fibrosis Level measured by KPa(kiloPascal) using SWE. F0 = Below 5 KPa, No fibrosis. F1=5.0-7.1 KPa, Mild Fibrosis. F2=7.1-8.7 KPa, Significant Fibrosis. F3=8.7-10.4 KPa, Sever Fibrosis. F4=10.4-19 KPa ,Cirrhosis. SWE can differentiate patients with no or minimal (F0 and F1) fibrosis from those with severe fibrosis or cirrhosis (F3 and F4) with no need for biopsy unless there are other factors that need to be considered.

SECONDARY OUTCOMES:
Shear Wave Elastography of spleen to asses spleen fibrosis in Gaucher disease patients. | 0-2 hours
  Shear wave elastography (SWE), an ultrasound imaging technique that can produce 2D and 3D images and quantified measurements of tissue stiffness noninvasively.
  Participants with Gaucher disease will under go shear wave elastography for spleen.
  Ultrasound Elastography is a non-invasive test which uses the technology of Shear Wave Elastography (SWE) obtained from the spleen for staging tissue fibrosis according to a study, Spleen Elastography was performed in 59 healthy individuals and the mean value measured in KPa (kiloPascal) was 16.6 ± 2.5 kPa, independent of patient age, sex or spleen size.
  above the normal value it is considerd fibrosis of the tisuue of the spleen.

OTHER OUTCOMES:
Biomarkers of the Gaucher Disease | Up to 1 month
  Gaucher Disease (GD) patients will be referred from the (GD) hematology outpatient clinic, in different patients different biomarker are already taken (as blood test).
  Biochemical abnormalities which might be already taken from patients, for example; blood level of ferritin (unit: ng/mL), angiotensin converting enzyme (unit: kU/L), chitotriosidase (unit: U/L) and polyclonal immunoglobulins (unit: ng/dL) .
  Elevated biomarkers can predict the severity of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: ziv neeman, MD, Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Northern District, Israel